CLINICAL TRIAL: NCT05029427
Title: Effect of Oat Beta Glucan in Managing Blood Pressure: a Randomized Cross-over Pilot Trial
Brief Title: Effect of Oat Beta Glucan in Managing Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Agriculture and Agri-Food Canada (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: HS24522(B2020:127)
Record Dates: First submitted 2021-08-26; First posted 2021-08-31 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Elevated Blood Pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Treatments will be provided to participants' homes via delivery. The treatments will be in similar looking breakfast cookies that will be prepared and delivered people outside of the clinical trial team.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study period 1: β-glucan Oat ; Study period 2: Wheat (Experimental): For the first period, the participant will receive food products made from oats containing a total of 4 grams per day HMW oat β-glucan. For the second period, the participant will receive food products made from wheat.
  Interventions: Other: High molecular weight β-glucan oat cookies; Other: Control wheat based cookies
- Study period 1: Wheat ; Study period 2: β-glucan Oat (Experimental): For the first period, the participant will receive food products made from wheat. For the second period, the participant will receive food products made from oats containing a total of 4 grams per day HMW oat β-glucan.
  Interventions: Other: High molecular weight β-glucan oat cookies; Other: Control wheat based cookies

INTERVENTIONS:
Other: High molecular weight β-glucan oat cookies — Two cookies that contains 4g beta glucan made from oats will be consumed per day.
Other: Control wheat based cookies — Two cookies that made from cream of wheat without beta glucan will be consumed per day.

SUMMARY:
This is a randomized, double-blinded, cross-over pilot study comparing the effects of ingesting oats containing high molecular weight β-glucan in reducing blood pressure.

DETAILED DESCRIPTION:
The pilot study will consist of 2 study periods: one treatment period and one control period. The treatment period will provide food products made from oats containing a total of 4 grams per day high molecular weight (HMW) oat β-glucan, whereas, the control period will provide food products made primarily from wheat with no β-glucan. The study will be located at the Chronic Disease Innovation Centre in Seven Oaks General Hospital, Winnipeg, Canada.

The primary objective of this study is to investigate the effect of ingestion of HMW oat β-glucan on ambulatory blood pressure. Participants will be asked to wear an ambulatory blood pressure monitor for 24 hours per day for 3 consecutive days at the beginning and end of each treatment period. This device automatically measures blood pressure every 15-30 minutes during the day and 30 to 60 minutes during the evening.

The study has been designed to be conducted virtually. Participants will consent to receive both treatment and control over two 4-week periods online. The participants will be randomized to different orders of treatment, with a 4 week wash out period in between.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the trial
* Generally healthy male and non-pregnant/lactating female, between the ages of 40-75
* When measured by the ambulatory blood pressure monitor, average systolic blood pressure (between 120 and 150mm Hg) and diastolic blood pressure (between 75 and 100mm Hg)
* Willing to comply with protocol requirements
* Willing to maintain their current weight and activity level throughout the study
* Body mass index 18.5-35kg/m2

Exclusion Criteria:

* Female participant who is pregnant, lactating or planning pregnancy during the course of the trial
* Body mass index ≤ 18.4 and ≥ 35.1 kg/m2
* If there is a history of a secondary cause of hypertension
* Ambulatory blood pressure monitor, systolic blood pressure >150mm Hg or <120mm Hg, diastolic pressure >100mm Hg or <75 mm Hg
* Use of medications containing pseudoephedrine or other vasoconstricting agents
* Antihypertensive drug treatment, regular high dose nonsteroidal anti-inflammatory drugs (NSAID) treatment and the use of cyclosporine or tacrolimus
* Cardiovascular disease including stroke, congestive heart failure, myocardial infarction, unstable angina pectoris, coronary artery bypass graft, percutaneous transluminal coronary angioplasty, temporal ischemic attack within six months prior to screening
* Not willing to maintain their regular physical activity level throughout the intervention
* Use of omega-3 fatty acid, herbal supplements or weight loss drugs
* Diagnosis of diabetes type 1 or type 2
* Scheduled elective surgery or other procedures requiring general anaesthesia during the trial
* Any other significant disease or disorder which, in the opinion of the Investigator or study physician, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial
* Recent history (within 6 month of screening) or current consumption of >14 drinks per week, (1 drink = 12oz of beer, 5oz of wine or 1.5oz distilled spirits)
* Body weight change over 3.5kg for the past 3 months
* Smokers and tobacco/snuff/nicotine users
* Allergy to oats, wheat, peanut, apple, cherry, blueberry, quinoa, egg white, margarine and vanilla extract.
* Regular consumption of supplements which may influence blood pressure/consumption of food supplements targeted to blood pressure lowering within 30 days before and during the study
* Participants who have participated in another research trial involving an investigational product in the past 12 weeks

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-11-28 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2022-12-23 (Actual)

PRIMARY OUTCOMES:
Mean systolic blood pressure | Day 1 to 3 and day 26-28 of each study period
  The mean systolic blood pressure will be measured for 24 hours for 3 consecutive days with an ambulatory blood pressure machine

SECONDARY OUTCOMES:
Body weight | Day 1 and day 28 of each study period
  Body weight will be measured in kg to the nearest 0.1 kg using a digital scale
Waist circumference | Day 1 and day 28 of each study period
  Waist circumference in cm will be measured in triplicate, to the nearest 0.1 cm at the umbilicus, between the last rib and iliac crest using a fibreglass tape
Mean diastolic blood pressure | Day 1, 2, and 3 and day 26, 27, and 28 of each study period
  The mean diastolic blood pressure will be measured for 24 hours for 3 consecutive days with an ambulatory blood pressure machine
Mean arterial blood pressure | Day 1, 2, and 3 and day 26, 27, and 28 of each study period
  The mean arterial blood pressure will be measured for 24 hours for 3 consecutive days with an ambulatory blood pressure machine

OTHER OUTCOMES:
Dietary fibre by 24 hour recall | Day 1, 2, and 3 and day 26, 27, and 28 of each study period
  Food recalls will be collected through Automated Self-Administered 24-hour dietary assessment tool and analyzed for consumption of dietary fibre

CONTACTS AND LOCATIONS:
Overall Officials: Dylan Mackay, PhD, Principal Investigator — University of Manitoba
Locations (1):
- Chronic Disease Innovation Centre, Seven Oaks Hospital, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) may be deposited in a repository if required by the journal where the results are published, otherwise it will be available upon request to the principle investigator.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: The data will be available following the publication of the primary results manuscript, and for a period of 25 years.
Access Criteria: Reasonable request to the principle investigator